CLINICAL TRIAL: NCT01471938
Title: Application and Adaption of Device Specific Body Composition Formulas to Various Ethnic Groups
Status: Completed | Type: Observational
Sponsor: Seca GmbH & Co. Kg. (Industry)
Responsible Party: Sponsor
Other Study IDs: BCA-02
Record Dates: First submitted 2011-07-08; First posted 2011-11-16 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2012-02

CONDITIONS: Bioelectrical Impedance Measurement of Healthy Adults

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Caucasians: 31 healthy adults in an age range of 18 to 65 years with a BMI of 18.5 to 35 kg/m2 are planned to be recruited.
- Afro Americans: 31 healthy adults in an age range of 18 to 65 years with a BMI of 18.5 to 35 kg/m2 are planned to be recruited.
- East and Southeast Asian: 31 healthy adults in an age range of 18 to 65 years with a BMI of 18.5 to 35 kg/m2 are planned to be recruited.
- Hispanics: 31 healthy adults in an age range of 18 to 65 years with a BMI of 18.5 to 35 kg/m2 are planned to be recruited.

SUMMARY:
The aim of the study is to apply and adapt device specific body composition formulas to various ethnic groups. Bases are prediction equations that are generated in the clinical investigation "Generation of prediction equation to analyze body composition of adults based on Bioelectrical Impedance Analysis (BIA)". The study bears the code BCA-01.

ELIGIBILITY:
Inclusion Criteria:

The study will cover 130 healthy adults. 65 men and 65 women in an age range of 18 to 65 years with a BMI of 18.5 to 35 kg/m2 are planned to be recruited.

Exclusion Criteria:

* acute and chronic diseases
* regular intake of medications (except for contraceptives)
* amputation of limbs
* electrical implant as cardiac pacemaker
* insulin pumps
* artificial joints
* metallic implants (except tooth implants)
* claustrophobia
* pregnancy or breastfeeding period
* probands who cannot provide an ICF by themselves
* probands who might be dependent from the sponsor or the inv. site
* current alcohol abuse
* frequent hypersensitivity reactions/allergies determ. anamnestically
* body weight of more than 150 kg
* extensive tattoos at arms or legs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Data of 130 healthy adults are planned to be collected.
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2011-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Bioelectrical Impedance (Resistance and Reactance) of 5 and 50 kHz for one body side | about 1 hour
Bioelectrical Impedance (Resistance and Reactance) of 50 kHz for all 4 extremities | about 1 hour
Bone Mineral Content (BMC) based on DXA (Dual X-Ray Absorptiometry) | about 30 minutes
  BMC is used to calculate Fat Free Mass (FFM). In addition to that Body Volume, Total Body Water (TBW) and Body Weight is needed. DXA is used as reference measurement for Skeletal Muscle Mass (SMM) as well.
Body Volume based on Air Displacement Plethysmography (ADP) | about 30 minutes
  Body Volume is used to calculate FFM in addition to DXA, TBW and Body Weight.
TBW | within 4 hours
  A D2O dose of 400 mg per kg body weight mixed with tap water is administered orally in the morning fasting and after a 2 hour fluid abstention. The distribution of the stable isotope in the TBW is completed after 4 hours. During this period, the subject remains fasting. Two venous blood samples of 10 ml whole blood are taken immediately before and four hours after taking D2O. The plasma samples are analyzed using Isoptopic Ratio Mass Spectrometry (IRMS).
ECW | within 4 hours
  Orally administered NaBr is resorbed quickly and completely and almost exclusively distributes in the extracellular compartment. Blood samples of 10 ml are taken immediately before and 4 hours after oral application of 50 mg NaBr per kg body weight. The serum sample is analyzed by X-Ray Fluorescence Spectroscopy (XRF).

SECONDARY OUTCOMES:
Bioelectrical Impedance (Resistance and Reactance) of 1, 1.5, 2, 3, 7.5, 10, 15, 20, 30, 75, 100, 150, 200, 300, 500, 750 and 1,000 kHz | about 1 hour
  The measurement is planned to be done for all body segments: right arm, left arm, right leg, left leg, trunk, right body side and left body side. In total resistance and reactance at 19 frequencies for 7 body segments are planned to be measured.
SMM based on Magnet Resonance Imaging (MRI) | about 1 hour
Bioelectrical Impedance (Resistance and Reactance) in sitting, lying and standing body position | about 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Dympna Gallagher, Dr., Principal Investigator — St. Luke's-Roosevelt Hospital Center
Locations (1):
- Body Composition of NY Obesity Research Center, New York, New York, United States

REFERENCES:
- [Derived] Jensen B, Braun W, Both M, Gallagher D, Clark P, Gonzalez DL, Kluckmann K, Bosy-Westphal A. Configuration of bioelectrical impedance measurements affects results for phase angle. Med Eng Phys. 2020 Oct;84:10-15. doi: 10.1016/j.medengphy.2020.07.021. Epub 2020 Jul 30. PMID 32977906